CLINICAL TRIAL: NCT03603262
Title: A Phase I, Open-label Study to Assess the Safety, Tolerability and Pharmacokinetics of Ascending Doses of SH-1028 Tablets in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Safety, Tolerability and Pharmacokinetics of SH-1028 in Patients With Advanced NSCLC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Sanhome Pharmaceutical, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHC013-I-01
Record Dates: First submitted 2018-07-04; First posted 2018-07-27 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2018-07

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — SH-1028

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SH-1028 (Experimental): Oral Once-Daily Administration of SH-1028
  Interventions: Drug: SH-1028

INTERVENTIONS:
Drug: SH-1028 — Starting dose 60mg,oral administered once daily.If tolerated subsequent cohorts will test increasing doses (100mg,200mg,300mg,400mg) of SH-1028.

SUMMARY:
This is a Phase 1, open-label study of SH-1028 with dose escalation and dose expansion cohorts in locally advanced or metastatic non-small-cell lung cancer (NSCLC) patients who have progressed following prior therapy with an epidermal growth factor receptor(EGFR) tyrosine kinase inhibitor (TKI) agent.

DETAILED DESCRIPTION:
The study is designed to evaluate safety, tolerability, pharmacokinetics (PK), and anti-tumor activity of once-daily and orally (PO) administered SH-1028 tablets. The overall study design is shown in the flow chart below, which consists of 2 phases: dose escalation and dose expansion cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 75, both sexes.
2. Histologically or cytologically documented NSCLC.
3. Not amenable to radical therapy or stage IV.
4. Radiological documentation of disease progression while on a previous continuous treatment with an EGFR TKI, e.g., gefitinib or erlotinib. In addition, other lines of therapy may have been given(chemotherapy only accept first line).
5. Confirmation that the tumor harbors an EGFR mutation known to be associated with EGFR TKI sensitivity (including G719X, exon 19 deletion, L858R, L861Q) or must have experienced clinical benefit from EGFR TKI, according to the Jackman criteria while on continuous treatment with an EGFR TKI(PR/CR、or SD continued ≥6 months).
6. Patients must have confirmation of tumor T790M+ mutation status.
7. Patients also must have confirmation of tumor T790M+ mutation status.
8. World Health Organization (WHO) performance status equal to 0-1 with no deterioration over the previous 2 weeks.
9. A minimum life expectancy of 12 weeks.
10. At least 1 lesion that has not previously been irradiated, that can be accurately measured at Baseline as ≥ 10mm in the longest diameter (except lymph nodes which must have short axis ≥ 15mm) with computerized tomography (CT) or magnetic resonance imaging (MRI), which is suitable for accurately repeated measurements.
11. Females of child-bearing potential should be using adequate contraceptive measures throughout the study, should not be breast feeding during the study and until 6 months after completion of study, and must have a negative pregnancy test prior to start of dosing.
12. Male patients should be willing to use barrier contraception during the study and until 6 months after completion of study (i.e., condoms).
13. Do not anticipate other clinical trail in 3 months.
14. The patient must provide a written informed consent for genetic research.

Exclusion Criteria:

1. Not Confirmed by pathology.
2. An EGFR TKI within 8 days or approximately 5 times the half-life of the specific drug, whichever is longer, of the first dose of study treatment.
3. Any cytotoxic chemotherapy used for a previous treatment regimen or clinical study within 21 days of the first dose of study treatment; Any target medicines used for a previous treatment regimen or clinical study within 14 days of the first dose of study treatment; withdrawal other clinical drugs or anti-cancer drugs less than 5 times the half-life.
4. Ever used the third EGFR-TKI, such as AZD9291,CO-1686 or avitinib.
5. Major surgery within 4 weeks of the first dose of study treatment.
6. Radiotherapy with a limited field of radiation for palliation within 1 week of the first dose of study treatment, with the exception of patients receiving radiation to more than 30% of the bone marrow or with a wide field of radiation which must be completed within 4 weeks of the first dose of study treatment.
7. The patient is currently using (or cannot discontinue at least 1 week before the first dose of study treatment) a drug or herbal supplement known as a potent inhibitor or inducer of CYP3A4.
8. Use large doses of glucocorticoids or other immunosuppressive agents within 4 weeks.
9. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE), Grade 1, at the time of starting study treatment with the exception of alopecia and Grade 2, prior platinum-therapy related neuropathy.
10. Spinal cord compression or brain metastases unless asymptomatic, stable, and not requiring steroids for at least 4 weeks prior to start of study treatment.
11. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension or active bleeding diatheses, which, in the Investigator's opinion, makes it undesirable for the patient to participate in the trial.
12. Active infection (e.g., hepatitis B, hepatitis C or human immunodeficiency virus [HIV]). (HBsAg is positive but HBV-DNA <1×103 IU/ mL ,and HCVAb is positive but HCV-RNA<103 IU/mL can be accepted.）.
13. Any of the following cardiac criteria:

    1. Mean resting corrected QT interval (QTc) > 470 msec obtained from 3 electrocardiograms (ECGs), using the Screening clinic ECG machine and Fridericia's formula for QT interval correction.
    2. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG (e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval >250msec).
    3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval.
14. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
15. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

    1. Absolute neutrophil count < 1.5 x 109/L.
    2. Platelet count < 100 x 109/L.
    3. Hemoglobin < 90 g/L (< 9 g/dL).
    4. Alanine aminotransferase > 2.5 times the upper limit of normal (ULN) if no demonstrable liver metastases or > 5 times the ULN in the presence of liver metastases.
    5. Aspartate aminotransferase > 2.5 times the ULN if no demonstrable liver metastases or > 5 times the ULN in the presence of liver metastases.
    6. Total bilirubin > 1.5 times the ULN if no liver metastases or > 3 times the ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases.
    7. Creatinine > 1.5 times the ULN concurrent with creatinine clearance < 50 mL/min (measured or calculated by the Cockcroft - Gault equation); confirmation of creatinine clearance is only required when creatinine is > 1.5 times the ULN.
16. Have any other malignant tumor within five years (except clinically cured cervical carcinoma in situ, basal cells or squamous epithelial skin cancer).
17. Refractory nausea, vomiting, or chronic gastrointestinal diseases, inability to swallow the study medication, or previous significant bowel resection that would preclude adequate absorption of SH-1028.
18. History of hypersensitivity to any active or inactive ingredient of SH-1028 or to a drug with a similar chemical structure or class to SH-1028.
19. Women who are breast feeding.
20. Any disease or condition that, in the opinion of the Investigator, would compromise the safety of the patient or interfere with study assessments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2018-04-25 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Within the first 28 days of treatment
Incidence of Dose Limiting Toxicity (DLT) | Within the first 28 days of treatment
Area under the plasma concentration versus time curve (AUC) of SH-1028 | 4 weeks
Elimination half-life(T1/2) of SH-1028 | 4 weeks
Maximum (or peak) concentration of SH-1028 | 4 weeks

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 12 months
Progression-free survival (PFS) | 12 months
Disease control rates（DCR） | 12 months
Overall survival（OS） | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: SHU YONGQIAN, MD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] He J, Ma P, Zhao D, Shi X, Guo R, Gao W, Shu Y. Safety, efficacy, and pharmacokinetics of SH-1028 in EGFR T790M-positive advanced non-small cell lung cancer patients: A dose-escalation phase 1 study. Cancer. 2023 May 15;129(10):1513-1522. doi: 10.1002/cncr.34697. Epub 2023 Feb 22. PMID 36813747